CLINICAL TRIAL: NCT01552265
Title: Shanghai Cohort Study on Mild Cognitive Impairment for Early Detection of Alzheimer's Disease
Brief Title: Shanghai Mild Cognitive Impairment Cohort Study
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: TRIAD1109
Record Dates: First submitted 2012-02-15; First posted 2012-03-13 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single-group MCI patients

SUMMARY:
This study was planned 1) to identify individuals with Mild Cognitive Impairment (MCI) who convert to Alzheimer's Disease (AD), and 2) to explore factors associated with the conversion.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive concern reflecting a change in cognition reported by the patient or informant or clinician
2. Mini-Mental State Examination (MMSE) scores between 18-30 (inclusive)
3. Clinical Dementia Rating (CDR) =0.5; Memory Box score must be at least 0.5
4. Objective memory loss* as evidenced by Auditory Verbal Learning test (AVLT-HS)
5. Essentially preserved activities of daily living based on Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
6. Not-demented, as defined by '"All-cause Dementia" (see 3.4. All-cause Dementia)
7. Willing to and able to undergo all test procedures including neuroimaging, and agree to longitudinal follow up
8. Written informed consent for the participation of this study including repeated neuropsychological tests and MRI scans

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-02; Primary Completion 2017-02 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Time to Conversion from MCI to "Probable AD Dementia" | 3 years

SECONDARY OUTCOMES:
Time to Conversion from MCI to "Possible AD Dementia" or "Probable AD Dementia" | 3 years
Time to Conversion from MCI to "All-cause Dementia" | 3 years
Overall survival | 3 years
Changes in Neuropsychological examinations | baseline, annual and 3 years
Changes in MRI | baseline, annual and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoji Nagai, MD,PhD, Study Director — Translational Research Informatics Center, Foundation for Biomedical Research and Innovation, Kobe,Japan
Locations (1):
- Department of Neurology, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou B, Zhao Q, Kojima S, Ding D, Higashide S, Nagai Y, Guo Q, Kagimura T, Fukushima M, Hong Z. One-year Outcome of Shanghai Mild Cognitive Impairment Cohort Study. Curr Alzheimer Res. 2019;16(2):156-165. doi: 10.2174/1567205016666181128151144. PMID 30484408
- See also: Related Info — http://www.tri-kobe.org